CLINICAL TRIAL: NCT06348992
Title: ACT (Acceptance Commitment Therapy) Combined with Yoga for Parental Burnout in Parents with Autistic Children: a Randomized Controlled Trial.
Brief Title: ACT Combined Yoga for Parental Burnout in Parents with Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Jiayi Chen, Principal Investigator, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HMUDQ20240318001
Record Dates: First submitted 2024-03-20; First posted 2024-04-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Parental burnout; Acceptance commitment therapy; Yoga; Psychosomatic intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acceptance and Commitment Therapy; Yoga

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT-Y (Experimental): Based on ACT and supplemented by Hatha Yoga exercise intervention, the intervention group used a combination of offline ACT psychological intervention and online Hatha Yoga training. ACT-Y intervention will be based on ACT combined with Yoga training and comprises a programme divided into eight 1-hour sessions conducted over 8 weeks
  Interventions: Behavioral: Acceptance commitment therapy and yoga
- Mental Health Education Group (Active Comparator): The control group also received 8 weeks of mental health education, including stress coping strategies, scientific parenting knowledge, and emotional management skills.
  Interventions: Behavioral: Active Comparator: Mental Health Education Group

INTERVENTIONS:
Behavioral: Acceptance commitment therapy and yoga — The intervention used a combination of online and offline methods, based on ACT, supplemented by hatha yoga exercise intervention, the intervention group used the combination of offline ACT psychological intervention and online hatha yoga training, and the control group used mental health education, so as to explore and validate the effect of ACT combined with yoga on the improvement of parental parental burnout in children with ASD. The offline ACT psychological intervention was implemented by the researchers and psychologists, and the ACT psychological intervention was carried out once a week in community health centers or hospitals for 8 weeks. Online, a WeChat group was set up for parents with ASD, and Hatha Yoga training content and videos were sent to the group chat, and the researchers and volunteers supervised the training and clocking in and out of the group, three times a week.
  Arms: ACT-Y
Behavioral: Active Comparator: Mental Health Education Group — The control group was provided with 8 weeks of mental health education, including emotional management skills, positive coping styles, and scientific parenting methods.
  Arms: Mental Health Education Group

SUMMARY:
OBJECTIVE: To explore the intervention effect of ACT combined with a yoga intervention program on parenting burnout in parents with ASD.

METHODS: This study used a combination of qualitative research and quantitative analysis to examine the intervention effects of an ACT-centered intervention program on parenting burnout in parents of children with ASD, and to clarify the evaluations and perceptions of parents with ASD about the research program through qualitative research.

RESULTS AND CONCLUSION: To clarify the intervention effect of ACT combined with yoga intervention program on parenting burnout of ASD parents.

DETAILED DESCRIPTION:
This study will focus on parents of children with ASD, and through literature review, intervention research, qualitative research, and other methods, based on PRO, adopt acceptance commitment therapy as the core intervention program to explore the improvement of parenting burnout, stress level and quality of life of parents, to enhance the psychological flexibility of parents with ASD, so that parents can positively cope with negative emotions and adverse events in life, and to promote the physical and mental health of parents and the quality of child care, so as to enhance the well-being and quality of life of families with ASD, and to enhance the well-being and quality of life of families with ASD. The program promotes the physical and mental health of parents and the quality of care for their children, thereby enhancing the well-being and quality of life of families with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children diagnosed with ASD based on DSM-5
* Parental burnout exists in parents
* Parents have normal speech, hearing and cognitive functioning
* Is the primary caregiver for children
* Informed consent and voluntary participation

Exclusion Criteria:

* Untreated ongoing or severe psychiatric disorders such as anxiety disorders, depressive disorders, schizophrenia, etc.;
* other more serious psychosomatic disorders that would interfere with the intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Measuring parental Burnout Levels | 3 months
  Developed by Roskam et al. to assess parenting burnout levels. There are 23 items in the scale, which are divided into four dimensions: the sense of exhaustion of the parental role, the boredom of the parental role, the emotional alienation from the children, and the self-comparison with the previous parental role. Scores range from 23-161. Higher scores indicate higher levels of parental burnout.
Measuring parenting stress Levels | 3 months
  The scale consists of 15 items divided into three dimensions: parenting distress (items 1-5), dysfunctional parent-child interactions (items 6-10), and difficult child characteristics (items 11-15). The total score ranges from 15 to 75, with higher scores indicating more severe parenting stress.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System adult profile-57, PROMIS-57 | 3 months
  VIII. Patient Self-Report PROMIS-57 This 57-item scale includes seven subscales on physical functioning (1-8 items), anxiety (9-16 items), depression (17-24 items), fatigue (25-32 items), sleep status (33-40 items), ability to assume social roles and participate in social activities (41-48 items), and the effects of pain (49-57 items).
Medical Outcomes Study 36-Item Short-Form Health Survey, MOS SF-36 | 3 months
  The scale, revised by Sun Yat-sen Medical University, is an internationally recognized universal quality of life evaluation scale with high reliability and validity. The scale has a total of 36 items, which are divided into 8 dimensions of quality of life, including physiological function, physiological function, physical pain, general health, vitality, social function, emotional function, and mental health.
Acceptance and Action Questionnaire-II, AAQ-II | 3 months
  The scale consists of 7 entries with a total score of 7-49, and the scores are summed so that the higher the score, the higher the level of empirical avoidance.
Cognitive Fusion Questionnaire，CFQ-F | 3 months
  Contains 9 entries with a total score of 9-63; the higher the total CFQ-F score, the higher the level of cognitive integration.

CONTACTS AND LOCATIONS:
Overall Officials: Quanzhi Zhang, Doctor, Study Chair — Harbin Medical University
Locations (1):
- Harbin Medical University Hospital, Daqing, None Selected, China

IPD SHARING:
Plan to Share IPD: No